## Different Conbercept Injection Methods in Treatment of Severe Proliferative Diabetic Retinopathy

NCT02816710 2016-06-30

## Statistical Analysis Plan

The results were analyzed using SPSS statistical software (version 19.0 for Windows, SPSS, Inc., Chicago, IL). Visual acuities were converted to logMAR before the statistical analysis. The Levene test was employed to assess the variance homogeneity of data distributions and the Kolmogorov-Smirnov test was employed to assure the normality of data distributions. The difference between groups were analyzed with chi-square test for categorical variables. One-way analysis of variance (ANOVA) was used for comparisons of normally distributed data, and Tukey's HSD test was used for comparisons of the differences between groups. For data that was not normally distributed, a Kruskal-Wallis test was used for data comparisons and a Mann Whitney U test was used for determination of the differences among the three groups. However, only the variables which were found to be statistically significant among the three groups were compared between each two groups. Sensitivities at fixed specificities (85% and 95%) were calculated for different parameters.